CLINICAL TRIAL: NCT01456325
Title: A Randomized, Phase III, Multicenter, Double-Blind, Placebo-Controlled Study Evaluating Efficacy and Safety of Onartuzumab (Metmab) in Combination With Tarceva (Erlotinib) in Patients With Met Diagnostic-Positive Non-Small Cell Lung Cancer Who Have Received Standard Chemotherapy for Advanced/Metastatic Disease
Brief Title: A Study of Onartuzumab (MetMAb) in Combination With Tarceva (Erlotinib) in Participants With Met Diagnostic-Positive Non-Small Cell Lung Cancer Who Have Received Chemotherapy For Advanced or Metastatic Disease (MetLung)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OAM4971g; GO27761 (Other: Hoffmann-La Roche); 2011-002224-40 (EudraCT Number)
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Erlotinib Hydrochloride; onartuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Onartuzumab+Erlotinib (Experimental): Participants will receive onartuzumab 15 milligrams per kilogram (mg/kg) intravenous (IV) infusion on Day 1 of every cycle of 3 weeks along with erlotinib 150 mg tablet orally once daily (QD) from Day 1, Cycle 1 until there is evidence of disease progression, death, or unacceptable toxicity, whichever occurred first.
  Interventions: Drug: Erlotinib; Drug: Onartuzumab (MetMab)
- Placebo+Erlotinib (Placebo Comparator): Participants will receive onartuzumab matching placebo on Day 1 of every cycle of 3 weeks along with erlotinib 150 mg tablet orally QD from Day 1, Cycle 1 until there is evidence of disease progression, death, or unacceptable toxicity, whichever occurred first.
  Interventions: Drug: Erlotinib; Drug: Placebo

INTERVENTIONS:
Drug: Erlotinib — Participants will receive erlotinib 150 mg tablet orally once daily from Day 1, Cycle 1.
  Other Names: Tarceva
Drug: Onartuzumab (MetMab) — Participants will receive onartuzumab 15 mg/kg IV infusion on Day 1 of every 3-week cycle.
  Other Names: RO5490258
  Arms: Onartuzumab+Erlotinib
Drug: Placebo — Participants will receive onartuzumab matching placebo on Day 1 of every 3-week cycle.
  Arms: Placebo+Erlotinib

SUMMARY:
This randomized, multicenter, double-blind, placebo-controlled study will evaluate the efficacy and safety of onartuzumab (MetMAb) in combination with Tarceva (erlotinib) in participants with incurable non-small cell lung cancer identified to be Met diagnostic-positive. Participants will be randomized to receive either onartuzumab (MetMAb) or placebo in combination with erlotinib. Anticipated time on study treatment is until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, greater than or equal to (>/=) 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Histologically or cytologically confirmed incurable Stage IIIb/IV NSCLC tumor
* Met diagnostic-positive status tested by immunohistochemistry (IHC)
* Results of endothelial growth factor receptor (EGFR)-activating mutation testing
* Radiographic evidence of disease
* Prior treatment with at least one platinum-based line of treatment (for stage IIIb/IV) and no more than one additional line of chemotherapy treatment; the last dose of chemotherapy must have been administered >/= 21 days prior to Day 1
* availability of tissue sample for diagnostic testing is required

Exclusion Criteria:

* More than 30 days of exposure to an investigational or marketed agent that can act by EGFR inhibition, or a known EGFR-related toxicity resulting in dose modifications (EGFR inhibitors including but not limited to gefitinib, erlotinib and cetuximab)
* Brain metastases or spinal cord compression not definitively treated with surgery and/or radiation, or previously treated central nervous system (CNS) metastases or spinal cord compression without evidence of stable disease for >/= 14 days
* History of another malignancy in the previous 3 years, unless cured by surgery alone and continuously disease free for at least 3 years; participants with prior history of non-invasive cancers are eligible
* Inadequate hematological, biochemical or organ function
* Significant history of cardiac disease
* Serious active infection at time of randomization or other serious underlying medical conditions that would impair the ability of the participant to receive protocol treatment
* Any inflammatory changes of the surface of the eye
* Clinically significant gastro-intestinal disease, including uncontrolled inflammatory gastro-intestinal diseases
* Pregnant or lactating women
* Positive for human immunodefinciency (HIV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2012-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Randomization until death (up to approximately 18 months) (assessed at the treating physician's discretion using the local standard-of-care practice)

SECONDARY OUTCOMES:
European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer Module (EORTC QLQ-LC13) Scores | Screening, Day 1 of Cycles 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22 (cycle length = 21 days), study drug discontinuation visit (up to approximately 18 months)
Onartuzumab Serum Concentrations | 1 hour pre-onartuzumab (Pr-O) infusion on Day 1 of Cycles 1, 2, and 4, 1 hour post-onartuzumab (Po-O) infusion on Day 1 of Cycle 1 (cycle length = 21 days and duration of infusion = 60 minutes), End of treatment (up to approximately 18 months)
Percentage of Participants With Disease Progression or Death | Randomization until disease progression or death, whichever occurred first (up to approximately 18 months) (assessed at the treating physician's discretion using the local standard-of-care practice)
Progression Free Survival (PFS) | Randomization until disease progression or death, whichever occurred first (up to approximately 18 months) (assessed at the treating physician's discretion using the local standard-of-care practice)
Percentage of Participants with an Objective Response Assessed Using RECIST V 1.1 | Randomization until disease progression or death, whichever occurred first (up to approximately 18 months) (assessed at the treating physician's discretion using the local standard-of-care practice)

CONTACTS AND LOCATIONS:
Overall Officials: Ivor Caro, M.D., Study Director — Genentech, Inc.
Locations (178):
- United States (50):
  - Chandler, Arizona
  - Hayward, California
  - Modesto, California
  - Oakland, California
  - Orange, California
  - Roseville, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - San Jose, California
  - Santa Clara, California
  - South San Francisco, California
  - Vallejo, California
  - Walnut Creek, California
  - Boca Raton, Florida
  - Clearwater, Florida
  - Fort Myers, Florida
  - Jacksonville, Florida
  - Chicago, Illinois
  - Urbana, Illinois
  - Bettendorf, Iowa
  - Sioux City, Iowa
  - Louisville, Kentucky
  - Annapolis, Maryland
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Ann Arbor, Michigan
  - Duluth, Minnesota
  - St Louis, Missouri
  - Omaha, Nebraska
  - Reno, Nevada
  - Farmington, New Mexico
  - Syracuse, New York
  - Chapel Hill, North Carolina
  - Canton, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Chattanooga, Tennessee
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Bristol, Virginia
  - Roanoke, Virginia
- Argentina (3):
  - La Plata
  - Quilmes
  - Santa Fe
- Australia (5):
  - Camperdown, New South Wales
  - Waratah, New South Wales
  - Chermside, Queensland
  - Adelaide, South Australia
  - Parkville, Victoria
- Belgium (5):
  - Brussels
  - Ghent
  - Gilly (Charleroi)
  - Liège
  - Namur
- Brazil (6):
  - Salvador/BA, Estado de Bahia
  - Lajeado, Rio Grande do Sul
  - Novo Hamburgo, Rio Grande do Sul
  - Jaú, São Paulo
  - São Paulo, São Paulo
  - Sorocaba, São Paulo
- Canada (4):
  - Saint John, New Brunswick
  - Sault Ste. Marie, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Chile (2):
  - Santiago
  - Temuco
- Croatia (4):
  - Čakovec
  - Dubrovnik
  - Pula
  - Zagreb
- France (11):
  - Besançon
  - Caen
  - Grenoble
  - Limoges
  - Marseille
  - Montpellier
  - Paris
  - Poitiers
  - Saint-Herblain
  - Suresnes
  - Vandœuvre-lès-Nancy
- Germany (12):
  - Bad Berka
  - Berlin
  - Großhansdorf
  - Hamburg
  - Heidelberg
  - Karlsruhe
  - Mainz
  - München
  - Oldenburg
  - Regensburg
  - Ulm
  - Villingen-Schwenningen
- Hong Kong (2):
  - Pokfulam
  - Shatin
- Hungary (3):
  - Edelény
  - Miskolc
  - Szombathely
- Ireland (2):
  - Cork
  - Dublin
- Israel (7):
  - Beersheba
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Ramat Gan
  - Rehovot
- Italy (9):
  - Aviano, Friuli Venezia Giulia
  - Genoa, Liguria
  - Milan, Lombardy
  - Monza, Lombardy
  - Rozzano, Lombardy
  - Orbassano, Piedmont
  - Ancona, The Marches
  - Lido di Camaiore, Tuscany
  - Perugia, Umbria
- Japan (14):
  - Aichi
  - Chiba
  - Ehime
  - Fukuoka
  - Hyōgo
  - Kanagawa
  - Kyoto
  - Miyagi
  - Okayama
  - Osaka
  - Saitama
  - Shizuoka
  - Tokyo
  - Yamaguchi
- Netherlands (3):
  - Amsterdam
  - Groningen
  - Maastricht
- Lima, Peru
- Poland (5):
  - Gdansk
  - Krakow
  - Lodz
  - Olsztyn
  - Poznan
- Russia (5):
  - Ivanovo
  - Krasnodar
  - Omsk
  - Saint Petersburg
  - Tomsk
- Serbia (2):
  - Belgrade
  - Kragujevac
- South Africa (3):
  - Bloemfontein
  - Johannesburg
  - Sandton
- South Korea (2):
  - Gyeonggi-do
  - Seoul
- Spain (5):
  - Barcelona, Barcelona
  - Sabadell, Barcelona
  - Madrid, Madrid
  - Seville, Sevilla
  - Valencia, Valencia
- Taiwan (3):
  - Changhua
  - Kaohsiung City
  - Taipei
- Ukraine (5):
  - Cherkassy
  - Chernivtsi
  - Dnipropetrovsk
  - Sumy
  - Zaporizhzhya
- United Kingdom (5):
  - Belfast
  - Grimsby
  - Leicester
  - London
  - Manchester

REFERENCES:
- [Derived] Koeppen H, Yu W, Zha J, Pandita A, Penuel E, Rangell L, Raja R, Mohan S, Patel R, Desai R, Fu L, Do A, Parab V, Xia X, Januario T, Louie SG, Filvaroff E, Shames DS, Wistuba I, Lipkind M, Huang J, Lazarov M, Ramakrishnan V, Amler L, Phan SC, Patel P, Peterson A, Yauch RL. Biomarker analyses from a placebo-controlled phase II study evaluating erlotinib+/-onartuzumab in advanced non-small cell lung cancer: MET expression levels are predictive of patient benefit. Clin Cancer Res. 2014 Sep 1;20(17):4488-98. doi: 10.1158/1078-0432.CCR-13-1836. Epub 2014 Mar 31. PMID 24687921